CLINICAL TRIAL: NCT05395234
Title: 'Cook Like A Boss' Online - an Investigation Into the Effectiveness of Conducting an Online Cooking 'Camp' Intervention
Brief Title: Cook Like A Boss Online: A Virtual One-week 'Camp-style' Cooking Intervention
Acronym: CLAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: University of Ulster (Other)
Responsible Party: Principal Investigator, Fiona Lavelle, Dr Fiona Lavelle, Postdoctoral Research Fellow, Queen's University, Belfast
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MHLS 21_24
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Perceptions, Self
Keywords: cooking; perceived motor competence; Childhood Wellbeing; Childhood Health; Children; Food Education

STUDY DESIGN:
Intervention Model Description: Cook Like A Boss Online is a single-group pre post intervention design
Masking Description: Masking was not possible due to the nature of the interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cook Like A Boss Online - virtual week long cooking camp (Experimental): The original Cook Like A Boss camp style intervention, was based on the Cook-Ed Model (Asher et al., 2020) and underpinned by SLT and ELT (Bandura & McClelland, 1977; Kolb, 1984). The content was developed to ensure it was age-appropriate in line with the guidelines (Dean et al., 2021a) and included co-creation. The camp was designed to introduce the children to a range of food and skills and to nurture an initial interest in cooking. The adapted online version of the camp included five daily videos of the original chef performing the recipes. Minor adaptions included the removal of cooking pasta from scratch due to equipment concerns, reordering the days, and chef suggestions around alternative equipment/ingredients to use. The five daily videos were: 1) Introduction & flatbreads; 2) Chicken Chowder; 3) Baking day; 4) Chilli non Carne; 5) Honey Chilli Chicken
  Interventions: Behavioral: Cook Like A Boss Online - virtual week long cooking camp

INTERVENTIONS:
Behavioral: Cook Like A Boss Online - virtual week long cooking camp — The original Cook Like A Boss camp style intervention, was based on the Cook-Ed Model (Asher et al., 2020) and underpinned by SLT and ELT (Bandura & McClelland, 1977; Kolb, 1984). The content was developed to ensure it was age-appropriate in line with the guidelines (Dean et al., 2021a) and included co-creation. The camp was designed to introduce the children to a range of food and skills and to nurture an initial interest in cooking. The adapted online version of the camp included five daily videos of the original chef performing the recipes. Minor adaptions included the removal of cooking pasta from scratch due to equipment concerns, reordering the days, and chef suggestions around alternative equipment/ingredients to use. The five daily videos were: 1) Introduction & flatbreads; 2) Chicken Chowder; 3) Baking day; 4) Chilli non Carne; 5) Honey Chilli Chicken

SUMMARY:
Cook Like A Boss Online is a public engaging virtual cooking camp styled intervention evaluating an adapted theory-driven co-created intervention designed to improve perceived cooking competence.

DETAILED DESCRIPTION:
Cook Like A Boss Online is a virtual cooking camp styled intervention, providing engaging virtual cooking activities for children to take part in safely from their homes during the COVID-19 pandemic. The online intervention is adapted from the original theory-driven, age-appropriate and co-created 'Cook Like A Boss' intervention (Dean et al., 2022), into daily cooking videos emailed to parents for children to cook along to, aiming to improve perceived cooking competence and wellbeing. Children aged 9-12 years will be recruited from across the island of Ireland (Republic of Ireland and Northern Ireland) to take part in the intervention. Due to the uncertainty of the pandemic and the need for the intervention to run five days consecutively (i.e. over a school holiday), it is deemed unethical to have a delayed intervention control group and all children will be provided the opportunity to take part in the intervention. Study outcomes include perceived cooking competence, perceived motor competence, wellbeing and process evaluation measures and will be collected at baseline and post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Within age range
* In primary school (before exposure to Home Economics)

Exclusion Criteria:

* Outside age range
* In secondary school

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 259 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Change in CooC11 (perceived cooking competence) score after 1 week intervention | Pre intervention to post intervention (1 week intervention)
  Validated measure of perceived cooking competence (Dean et al., 2021b), completed by children. CooC11 is an 11-item measure used to assess children aged 8-12 years on their perceived competence of their cooking skills, including skills such as chopping, peeling, weighing ingredients and using an oven. Children are shown illustrations of characters and asked whether they do the skill, if they respond yes, they are then shown two illustrations one of a 'good' performance of a skill and one of a 'poor' performance. The child is then asked which image they are most like on a five point Likert scale. The sequence of presentation of 'good' and 'poor' performance of a skill alternated, and scores were reverse coded where necessary so that a higher score indicated a higher perceived competence. The score for each skill is then summed to create a total cooking competence score, with possible scores ranging from 0 to 55.
Change in perceived motor competence score after 1 week intervention | Pre intervention to post intervention (1 week intervention)
  Validated measure of perceived motor competence (Barnett et al., 2015), completed by the children. This is a 12-item measure, where children are shown images of children performing different physical activities and asked to pick which child they are like.
Change in Stirling Children's Wellbeing Scale score after 1 week intervention | Pre intervention to post intervention (1 week intervention)
  Validated measure of wellbeing (Liddle and Carter, 2015), completed by the children. This is a 15-item measure, where children select one of the following responses for the 15-items: 'Never,' 'Not much of the time,' 'Some of the time,' 'Quite a lot of the time,' 'All of the time.'

SECONDARY OUTCOMES:
Process evaluation measures | Pre to Post intervention (1 week intervention)
  Both parents and children answered a number of questions relating to their experiences of camp. Parents completed questions relating to the number of videos completed, rating their child's experience of camp, would they encourage their children to take part in more cooking activities in the home, surprise around children's abilities, changes in their children's cooking confidence. Children completed questions relating to enjoyment of camp, whether they would take part again, favourite part of camp, and what they learnt in camp.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Lavelle, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Institute for Global Food Security, Queen's University Belfast, Belfast, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hollywood L, Issartel J, Gaul D, McCloat A, Mooney E, Collins CE, Lavelle F. Cook like a Boss Online: an adapted intervention during the COVID-19 pandemic that effectively improved children's perceived cooking competence, movement competence and wellbeing. Int J Behav Nutr Phys Act. 2022 Dec 9;19(1):146. doi: 10.1186/s12966-022-01378-x. PMID 36494840